CLINICAL TRIAL: NCT04514406
Title: APERTO CVS PMCF Study: Drug Coated High Pressure Balloon in Large Veins (re)Stenosis in Dialysis Patients
Brief Title: APERTO CVS PMCF Study
Acronym: APERTO CVS
Status: Terminated | Type: Observational
Why Stopped: no enrolments
Sponsor: Cardionovum GmbH (Industry)
Collaborators: CliPS Service (Unknown); OPIS srl (Unknown)
Responsible Party: Sponsor
Other Study IDs: APERTO CVS
Record Dates: First submitted 2020-08-05; First posted 2020-08-17 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Dialysis; Complications; Central Vein Obstruction; Stenosis; Restenosis
Keywords: Drug Coated Balloon; Central Veins Stenosis; Percutaneous Intervention
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- APERTO OTW DCB: Dialysis patients treated with APERTO OTW following (re)stenosis of central veins
  Interventions: Device: APERTO OTW DCB

INTERVENTIONS:
Device: APERTO OTW DCB — Drug Coated Balloon Angioplasty

SUMMARY:
Prospective Observational Single Arm study aimed to assess safety and effectiveness of APERTO OTW DCB in treating stenosis and restenosis of central veins in dialysis patients

DETAILED DESCRIPTION:
The APERTO CVS PMCF study is aimed to evaluate safety and effectiveness of treatment of central veins (re)stenosis in dialysis patients at short and mid-term follow up, after treatment with APERTO OTW DCB. Primary endpoint will consist in evaluating the intervention free period for patients treated with APERTO OTW.

APERTO CVS PMCF Study will also collect data for post-market clinical follow up (PMCF) in a CE mark device used according to intended use

ELIGIBILITY:
Inclusion Criteria:

* Patients age >18, no pregnant women, able to perform fup visits, life expectancy > 12 months
* Dialysis patients undergoing endovascular angioplasty due to clinically symptomatic stenosis (de novo or restenosis) of the central veins with significant (>50%) stenosis and diameter
* The target lesion consists of one or more lesions with a target lesion length of less than or equal to 100 mm
* The target blood vessel diameter of the target lesion is between 6.0 and 16.0 mm (in angiographic or ultrasound evaluation);
* If there are other non-target lesions, then non-target lesions must be successfully cured with a not drug coated balloon before treating the target lesion;

Exclusion Criteria:

* Patients with CVS observed and estimated as nonsignificant (< 50% stenosis) or a vessel > 12 mm in diameter by visual estimation;
* the patient is now participating in another clinical trial to evaluate drug or medical device;
* patient enrolled for this trial before;
* prenatal pregnancy test result for women of childbearing potential is non-negative, Lactating woman;
* patients, who underwent major surgical procedures (such as thoracotomy, craniotomy, etc.) within 30 days prior to the study;
* patients scheduled to undergo major surgery (eg, thoracotomy, craniotomy, etc.) within 30 days after enrolment;
* central veins lesions have been already treated with DCB before
* presence of a bare metal stent (BMS) or stent graft or vascular access thrombosis in central veins
* patients allergic or intolerant to paclitaxel, or contrast media;
* patients whose life expectancy is less than 1 year
* presence of Thrombus in central veins
* tumor compression
* thoracic inlet syndrome
* patients implanted with pacing or cardioverter devices with leads
* any other central line within the target lesion
* Patients with any contraindications as mentioned in the Instructions for Use (IFU) of the Investigational Device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dialysis patients with symptoms for stenosis or restenosis of central veins to be treated with percutaneous angioplasty.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Clinically Assessed Intervention free period at 6 months fup | 6 months
  clinically assessed intervention free period at 6 months (IFP) defined as dialysis access circuit with no need for clinically driven target lesion repeat intervention for symptom recurrence

SECONDARY OUTCOMES:
Procedural Technical Success | intraoperative
  Residual stenosis is no more than 30% after treatment with APERTO OTW measured by angiography
Procedural Clinical Success | intraoperative
  After the procedure, haemodialysis access function improved, dialysis function restored, and at least one dialysis session completed
Procedural Surgical Success | intraoperative
  On the basis of technical success, no major adverse events (MAE) occurred during hospitalization or treatment
Major Adverse Event | 12 months follow up
  include death, stroke, thrombosis, allergic reactions, and pulmonary diseases (including pulmonary edema), bleeding complication with the need of transfusion
Fistula Flow | 6 months
  Flow measured with Echo Doppler measured at 6 months
Recirculation Rate | 6 months
  Recirculation rate measured at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Petra Michel, MD, Principal Investigator — Klinikum Hochsauerland; Michael Lichtenberg, MD, FESC, Study Director — Klinikum Hochsauerland
Locations (2):
- Germany (2):
  - Vivantes Klinikum, Berlin
  - St.Franziskus Hospital, Münster

IPD SHARING:
Plan to Share IPD: No